CLINICAL TRIAL: NCT05890573
Title: Efficacy of Bailing Capsule on Pulmonary Fibrosis After COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0091
Record Dates: First submitted 2023-05-29; First posted 2023-06-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Fibrosis; COVID-19 Pneumonia
Keywords: PCPF; COVID-19; Bailing Capsule
MeSH Terms: conditions — Pulmonary Fibrosis; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bailing capsule group (Experimental): Bailing capsule group:6 Bailing capsules,po, tid,12 weeks.
  Interventions: Drug: Bailing capsule
- Blank group (No Intervention): Blank group:no anti-fibrosis treatment is given.

INTERVENTIONS:
Drug: Bailing capsule — 6 Bailing capsules,po,tid,12 weeks
  Arms: Bailing capsule group

SUMMARY:
Pulmonary fibrosis is a sequela of severe infection COVID-19.The prevalence of PCFP ranged from 2% to 45%,and the pathogenesis of PCFP has not been clearly elucidated.The ingredient of Bailing capsule is Cs-C-Q80,it has obvious protective effect on lung.

Studies have shown that Bailing capsule may improve the clinical symptoms of PCPF patients through anti-fibrosis, oxidation and anti-inflammatory effects in multiple pathways.

The purpose of this study was to evaluate the efficacy and safety of bailing capsule in treating PCFP after COVID-19 infection.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open, randomized controlled clinical study. Bailing capsule was used for 12 weeks of convalescent treatment in patients with COVID-19 infection to evaluate the efficacy and safety of Bailing capsule on pulmonary fibrosis changes after COVID-19 infection.

The study consisted of a 1-week screening period and a 12-week randomized treatment period.

Screening period (V0) :

All subjects who have signed informed consent will enter a screening period (up to 7 days) to assess eligibility. Subjects with confirmed pulmonary fibrosis changes after COVID-19 infection were required to complete relevant procedures, examinations and assessments according to the study procedure table during the screening period.

Randomized treatment period (V1~V3) :

The randomized treatment period included V1 to V3 visits. At baseline visit (V1), eligible subjects will be randomly assigned to 6 capsules of Bailing Capsule, tid group, or blank control group in a 1:1 ratio, and receive appropriate treatment during the treatment period:

1. Experimental group: 6 capsules of Bailing capsule, tid group (n=121), a total of 12 weeks.
2. Control group: blank control (n=121).

During randomized treatment, subjects will be required to complete procedures, examinations, and evaluations according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old, gender unlimited;
2. Fibrous changes in the lungs after COVID-19 pneumonia:

   1. If COVID-19 is positive within the past 2 months, qualitative analysis of SARS-CoV-2 RNA is conducted by antigen detection or PCR detection;
   2. During the screening period, chest HRCT showed the characteristics of pulmonary interstitial lesions (including ground glass shadow, grid shadow, tractable bronchiectasis, septal thickening and early honeycomb shadow, etc.), with fibrosis affected area > 5%;
   3. COVID-19 negative was confirmed during the screening period, and SARS-CoV-2 RNA was qualitatively verified by antigen detection or PCR detection;
3. Severity grade 2 (moderate) or 3 (severe) according to the mMRC Dyspnea Scale at the screening visit;
4. Able to perform pulmonary function tests (PFT) and decreased lung function FVC and/or DLCO <70% of the predicted value at the screening visit;
5. Able to complete the 6-minute walking test and questionnaire survey;
6. Fertile female patients must have negative pregnancy test results during screening;
7. Volunteer to participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Prior medical history of lung disease (including IPF, bronchial asthma, COPD, lung cancer or pulmonary hypertension) prior to positive diagnosis of COVID-19 pneumonia;
2. Nephrotic syndrome, moderate to severe chronic renal failure, or eGFR < 60ml/min at enrollment;
3. Major cardiovascular disease, including chronic heart failure grade III or IV, clinically significant sinus arrhythmias, ventricular tachycardia, ventricular fibrillation, unstable angina, and severe hypertension (≥160/110 mmHg) that was not under control or was being actively treated within the first 6 months of enrollment;
4. Screening of patients with abnormal liver function, the criteria are as follows: total bilirubin > 1.5×ULN; ALT > 3 x ULN; AST > 3 x ULN;
5. Severe pulmonary arterial hypertension (PAH) meets any of the following conditions:

   1. severe right heart failure in the past;
   2. Cardiac index indicated by right cardiac catheter insertion history ≤2 L/min/m²;
   3. PAH requiring epizoprostol/treprostol parenteral treatment;
6. Patients with bleeding risk:

   1. Known genetic susceptibility to bleeding;
   2. fibrinolysis, full-dose anticoagulant therapy, or high-dose antiplatelet therapy are required;
7. Patients had received chest and neck radiotherapy or chemotherapy before screening;
8. Inability to swallow the study drug;
9. History of active malabsorption disorders or gastrointestinal resection;
10. Systemic corticosteroids (e.g. Prednisone, dexamethasone) were administered within 5 days of the first day of administration of the study intervention;
11. After discharge, take preparations containing cordyceps or anti-pulmonary fibrosis drugs (such as pirfenidone, Nidanib, imatinib, penicillamine, colchicine, tumor necrosis factor α receptor blockers, etc.);
12. Participation in other clinical trials, use of other investigational drugs or investigational devices within 30 days prior to randomization;
13. Women or men of childbearing age refuse to use contraception during the study period;
14. Pregnant or lactating women;
15. Any other factors that the investigator has determined may be inappropriate for participation in the clinical study;
16. Patients suffered major trauma or underwent major surgery within 28 days prior to treatment with the study drug;
17. Other Chinese medicines containing cordyceps were used for treatment within 15 days before and during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2024-04-16 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of clinically significant change in FVC and/or DLCO at Week 12 relative to the baseline value | Week 12
  Clinically significant changes include a relative ≥ 10% increase in FVC or a relative increase in FVC within the range from ≥ 5% to <10% and a relative ≥ 15% in DLCO

SECONDARY OUTCOMES:
Change in distance covered for 6 minutes (6MWD) from the baseline value (based on 6-minute walk test) | Week 4，Week 8，Week 12
  6MWD changing value
FVC | Week 4，Week 8，Week 12
  FVC（L）changing value
DLCO | Week 4，Week 8，Week 12
  DLCO（ mmHg）changing value
FEV1 | Week 4，Week 8，Week 12
  FEV1（ L）changing value
FEV1/FVC | Week 4，Week 8，Week 12
  FEV1/FVC（ %）changing value
TLC | Week 4，Week 8，Week 12
  TLC（ L）changing value
The rate of reduction in the lung damage degree based on the high-resolution computed tomography(HRCT) at Week 12 relative to the baseline value | Week 12
  Classification of lung damage includes the following stages: CT-0 (norm), CT-1 (< 25% of lung damage), CT-2 (25-50% of lung damage), CT-3 (50-75% of lung damage), CT-4 (> 75% of lung damage)
Change in mMRC Dyspnea Score from the baseline value | Week 12
  m-MRC changing value
Change in the overall score of the SF-36 Questionnaire relative to the baseline value | Week 12
  36-item Short-Form（SF-36） is a universal scale of life quality developed by Medical Outcomes Study（MOS）, which is widely recognized and used in the world. This scale has 8 dimensions to evaluate health-related quality of life (HRQOL), which can be divided into two categories of physiological health and mental health, namely physiological function (PF), role-physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role-emotional (RE) and mental health (MH). 50 is a normal average score, 0 is the lowest, 100 is the highest.The higher the score, the better the health.
Change in the overall score of the CQ-11D Questionnaire relative to the baseline value | Week 12
  TCM Life Quality Evaluation Scale (CQ-11D) is an industry standard document approved and officially released by the China Association of Traditional Chinese Medicine. It is mainly used to evaluate the healthy life quality of the population receiving TCM intervention and the general population, with a total of 11 items. The higher the score, the worse the healthy quality of life status.
The rate of adverse events (AEs) | Week 4，Week 8，Week 12
  AE

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Dai, Professor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Dai Haibin, Hangzhou, Zhejiang, China